CLINICAL TRIAL: NCT07348380
Title: Volatile Organic Compounds Analysis for Rapid Testing Using EXhaled Breath for Respiratory Infection
Brief Title: Volatile Organic Compounds Analysis by PTR-TOF-MS for Screening Respiratory Infections Using Exhaled Breath.
Acronym: VORTEX 1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL25-0599; 2025-A01542-47 (Other: ID-RCB)
Record Dates: First submitted 2025-11-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Infections; Respiratory Infections, Acute
Keywords: Pandemic preparedness; Volatilome; Breath research
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional diagnostic study using case-control sampling, where the number of cases and non-cases is fixed in advance, and a gold standard comparison is used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bacterial respiratory infection (Experimental): To classify patients, an adjudication committee will base its decision on a range of clinical and biological factors:
  * The ICD-10 code (International Classification of Diseases, 10th revision) assigned to the patient during their treatment
  * Radiological examination indicating bacterial pneumonia (community-acquired pneumonia or CAP)
  * Biological results:
    * Microbiological diagnostic tools (RT-PCR tests, culture) indicating a bacterial infection.
    * Procalcitonin measurement (indicating a bacterial infection if > 0.1 µg/L)
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using PTR-TOF-MS
- Viral respiratory infection (Experimental): To classify patients, an adjudication committee will base its decision on a range of clinical and biological factors:
  * The ICD-10 code (International Classification of Diseases, 10th revision) assigned to the patient during their treatment
  * Radiological examination not indicating bacterial pneumonia
  * Biological results:
    * Microbiological diagnostic tools (RT-PCR tests, culture) indicating a viral infection. For example, respiratory infections will be attributed to a virus if at least one of the diagnostic tests used is positive for a virus or if the interferon test shows a very high score.
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using PTR-TOF-MS
- Undetermined respiratory infection (Experimental): All patients who matched the inclusion criteria and could not be classified into groups 1 or 2 by an adjudication committee.
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using PTR-TOF-MS
- Healthy patients (Placebo Comparator): The group of healthy volunteers, serving as the control group, will be composed of adult subjects with no respiratory symptoms or known acute or chronic pathology at the time of inclusion. They will be sampled using the same methods as the other groups in order to enable a reliable comparison of the metabolic signatures obtained.
  Interventions: Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using PTR-TOF-MS

INTERVENTIONS:
Device: Volatile Organic compounds (VOC) analysis in Exhaled breath using PTR-TOF-MS — The collection and analysis of exhaled air for VOC detection is a non-invasive, painless procedure that will be carried out online and summarised as follows: . The patient's exhaled air is collected directly in the analyzer using disposable mouthpieces.
  2. Real-time chemical analysis of exhaled air over a few seconds (breath duration) using PTR-TOF-MS.
  3. Processing raw data to establish the chemical composition of VOCs. 4. Statistical analysis of all generated data to identify specific VOC profiles.
  Results will be compared to standard diagnostic procedure and linked to immune, metabolic and microbiome exploration.

SUMMARY:
Emerging respiratory diseases are a global health threat. Viruses such as influenza and coronaviruses have been the main cause of pandemics over the last century. In general, the impact of these respiratory infections is not limited to pandemic risks. Indeed, some pathogens also induce seasonal epidemics with a significant medical and economic burden. It is therefore essential to strengthen global surveillance, warning systems and early diagnosis capabilities for pathogens responsible for respiratory infections.

One promising and recognized approach is the analysis of exhaled air, which contains a complex mixture of volatile organic compounds (VOCs), also known as the "volatilome".

The volatilome is influenced by the patient's metabolism, immune system and microbiome. It can be disturbed by the presence of a pathogen.

A possible approach to study the human volatilome is called the "on-line" method. Among the technologies capable of performing online analysis, analyzers using TOF (time-of-flight) technology separate ions according to velocity differences after acceleration by a fixed potential, and then measure all mass/charge ratios simultaneously. The data obtained takes the form of a mass spectrum composed of a multitude of peaks representing the abundance of each detected chemical species contained in the exhalation. The sensitivity and measurement speed of instruments using PTR-TOF-MS (Proton Transfer Reaction - Time of Flight - Mass spectrometer) technology enable real-time monitoring of the exhalation process, making it possible to analyze exhaled air as a function of time. PTR-TOF-MS instruments are usually compact in design, enabling them to be deployed in environments such as hospital emergency wards or mass screening centers.

The aim of the VORTEX-1 study is to include patients presenting with signssymptoms of respiratory infections, irrespective of microbiological etiology, to approximate a routine clinical context, thus including infections of various viral or bacterial origins. In addition, a so-called "control" group will also be sampled, made up ofcomposed by healthy subjects (with nowithout respiratory infections or serious or chronic pathologies at the time of sampling).

In parallel with the study of the chemical composition of the exhaled air of these patients, and to further our understanding of the factors influencing the volatilome, a combined exploratory analysis of the respiratory microbiota, the host response at the time of infection, and the pathogen(s) responsible for the infectious episode is required. To date, no such analysis exists in the scientific literature, probably due to the technical and logistical complexity of integrating data from multiple sources and the lack of a multidisciplinary consortium with the necessary expertise.In parallel with the study of the chemical composition of the exhaled air of these patients, and in order to go further in understanding the factors influencing the volatilome, a combined exploratory analysis of the respiratory microbiota, the host response at the time of infection and the pathogen(s) responsible for the infectious episode is required. To date, no such analysis exists in the scientific literature, probably due to the technical and logistical complexity of integrating data from multiple sources, but also to the absence of a multidisciplinary consortium capable of bringing together all the necessary expertise within the same project.

The detection of specific VOCs could considerably improve and facilitate the diagnosis of these respiratory diseasesinfections.

This research could revolutionize the diagnosis of respiratory infections by offering a rapid, non-invasive and easily scalable alternative to conventional diagnostic methods such as PCR tests, which require nasopharyngeal sampling. In parallel with the study of the chemical composition of the exhaled air of these patients, and to further our understanding of the factors influencing the volatilome, a combined exploratory analysis of the respiratory microbiota, the host response at the time of infection, and the pathogen(s) responsible for the infectious episode is required. To date, no such analysis exists in the scientific literature, probably due to the technical and logistical complexity of integrating data from multiple sources and the lack of a multidisciplinary consortium with the necessary expertise.

The detection of specific VOCs could considerably improve and facilitate the diagnosis of these respiratory infections. by offering a rapid, non-invasive and easily scalable alternative to conventional diagnostic methods such as PCR tests.

ELIGIBILITY:
Eligibility Criteria *

* Inclusion Criteria * :

  * Age ≥ 18 years old
  * Having signed a written informed consent
  * With clinical signs of acute respiratory infection, or with a clinical presentation of acute community-acquired pneumonia, nasopharyngitis, angina or laryngitis (except for healthy patients)
* Exclusion Criteria * :

  * Healthy volunteers:
  * Age: < 18 years
  * Alcohol consumption less than 12 hours
  * Person with co-morbidities such as chronic respiratory failure, type II diabetes, cancerous processes, chronic liver disease, chronic kidney disease
  * Clinical signs of acute respiratory infection
  * Persons who are unable to blow into exhaled-air analysis devices (in accordance with instructions for use)
  * Persons under legal protection
  * Pregnant women, women in labor or nursing mothers
  * Persons deprived of their liberty by judicial or administrative decision
  * Persons under psychiatric care
  * Persons admitted to a health or social institution for purposes other than research
  * Adults under legal protection (guardianship, curatorship)
  * Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
  * Patients with respiratory symptoms
  * Age: < 18 years
  * Patients whose symptoms have been present for more than 7 days
  * Persons unable to blow into the device for breath analysis (in accordance with the operating instructions)
  * Patients suffering from cystic fibrosis
  * Patients with severe chronic respiratory insufficiency requiring long-term oxygen therapy or NIV (non-invasive ventilation), excluding CPAP (Continuous Positive Airway Pressure) for sleep apnea
  * Patients under legal protection
  * Pregnant women, women in labor or nursing mothers
  * Persons deprived of their liberty by judicial or administrative decision
  * Persons under psychiatric care
  * Persons admitted to a health or social institution for purposes other than research
  * Adults under legal protection (guardianship, curatorship)
  * Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1665 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-02 (Estimated)

PRIMARY OUTCOMES:
Comparison and differentiation between patients presenting symptoms of acute respiratory infection (ARI) and a control group of healthy subjects | DAY 1
  The test will aim to differentiate patients with one of the symptoms of acute respiratory infection from the control group of healthy patients. The overall performance of the test will be evaluated on several models, based on the area under the ROC curve (AUC) calculated from model predictions. Predicted AUCs will be compared to an expected AUC of 0.7 by bootstrapping.

SECONDARY OUTCOMES:
Validation of descriptive analyses of exhaled air test based on aggregated diagnostic parameters compared with those of the current biological reference standard for respiratory infection. | DAY 1
  Evaluate the performance (same as main objective) of the chemical analysis of exhaled air in differentiating between three groups of participants: those with a respiratory infection caused by a virus, those with a respiratory infection caused by bacteria, and healthy subjects.
Description of the breath composition based on the area under each peak of exhaled air according to six levels of classification | DAY 1
  Evaluate the performance of chemical analysis of exhaled air in differentiating between the following six groups of patients:
  * respiratory infection with Legionella spp.
  * respiratory infection with another bacterium
  * respiratory infection with SARS-CoV-2
  * respiratory infection with influenza
  * respiratory infection with another virus
  * uninfected patients
Description of the breath composition based on the AUC of each peak | DAY 1
  Analyse and describe the composition of patients' exhaled air according to viral (influenza and SARS-CoV-2) or bacterial (Legionella) load, in order to identify biomarkers whose excretion correlates with viral and bacterial load.
Description of the breath composition based on the AUC of each peak | DAY 1
  Analyse and describe the composition of patients' exhaled air based on the presence of co-infection, in order to define biomarkers whose excretion is associated with these co-infections.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre GAYMARD, MD, Principal Investigator — Centre National de Référence des virus des infections respiratoires Laboratoire de virologie Institut des Agents Infectieux
Locations (3):
- France (3):
  - Emergency department (Hôpital de la Croix-Rousse, Hospices Civils de Lyon) Lyon (France) 69004, Lyon
  - Maison de Santé Pluriprofessionnelle Universitaire (Hôpital de la Croix-Rousse, Hospices Civils de Lyon), Lyon
  - National reference center for respiratory viruses (Hôpital de la Croix-Rousse, Hospices Civils de Lyon), Lyon

IPD SHARING:
Plan to Share IPD: No